CLINICAL TRIAL: NCT05766865
Title: Effect and Safety of Surgical Intervention for Severe Spontaneous Intracerebral Hemorrhage Patients on Long-term Oral Antiplatelet Treatment
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Shuyi Hospital (Other); Beijing Anzhen Hospital (Other); Guangzhou Red Cross Hospital (Other); Beijing Pinggu District Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: KY2019-096-02
Record Dates: First submitted 2022-11-23; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Severe Spontaneous Intracranial Hemorrhage; Long-term Antiplatelet Treatment; Emergency Surgery; Complications
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency neurosurgery — Surgical evacuation for intracerebral hemorrhage
Procedure: Conservative treatment — Standard treatment for intracerebral hemorrhage

SUMMARY:
Background: Despite the capability of emergency surgery to reduce the mortality of severe spontaneous intracranial hemorrhage (SSICH) patients, the effect and safety of surgical treatment for severe spontaneous intracranial hemorrhage (SSICH) patients receiving long-term oral antiplatelet treatment (LOAPT) remains unclear. In consideration of this, the cohort study is aimed at figuring out the effect and safety of emergency surgery for SSICH patients on LOAPT.

Methods: As a multicenter and prospective cohort study, it will be conducted across 7 representative clinical centers. Starting in September 2019, the observation is scheduled to be completed by December 2022, with a total of 450 SSIC H patients recruited. The information on clinical, radiological, and laboratory practices will be recorded objectively. All of the patients will be monitored until death or 6 months after the occurrence of primary hemorrhage.

Results: In this study, two comparative cohorts and an observational cohort will be set up. The primary outcome is the effect of emergency surgery, which is subject to assessment using the total mortality and comparison in the survival rate of SSICH patients on LOAPT between surgical treatment and conservative treatment. The second outcome is the safety of surgery, with the postoperative hemorrhagic complication which is compared between the operated SSICH patients on and not on LOAPT. Based on the observation of the characteristics and outcome of SSICH patients on LOAPT, the ischemic events after discontinuing LOAPT will be further addressed, and the coagulation function assessment system for operated SSICH patients on LOAPT will be established.

Conclusions: In this study, we will investigate the effect and safety of emergency surgery for SSICH patients on LOAPT, which will provide an evidence for management in the future.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18-75 years old;
* (2) non-traumatic intracerebral hemorrhage;
* (3) severe intracerebral hemorrhage, which was defined as patients with supratentorial bleeding volume > 30 ml, infratentorial bleeding volume > 10 ml, midline shift > 1 cm, or large intraventricular hematoma;
* (4) Glasgow coma score (GCS) < 13;
* (5) family members agree to provide an informed written consent.

Exclusion Criteria:

* (1) patients had cerebrovascular diseases, e.g., intracranial aneurysm or vascular malformation, and intracranial tumors, which were associated with hemorrhage;
* (2) hemorrhagic transformation of cerebral infarction;
* (3) hemorrhage caused by venous thrombosis;
* (4) patients with severe coagulation disorder, e.g., hemophilia;
* (5) patients with coagulation dysfunction caused by malignant tumor, hepatic insufficiency, renal dysfunction, thrombocytopenia, coagulation diseases, and so on;
* (6) patients receiving other anticoagulation medications (vitamin K antagonist and new oral anticoagulants);
* (7) patients not on LOAPT who receive conservative treatment;
* (8) the patients who died before or on arriving at the hospital and within a short period (6 h) after admission.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All severe spontaneous intracerebral hemorrhage (SSICH) patients except those not on long-term oral antiplatelet treatment (LOAPT) receiving conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Total mortality | From admission to 6 months after the occurrence primary hemorrhage

SECONDARY OUTCOMES:
Postoperative intracranial bleeding | Within one week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordonnier C, Demchuk A, Ziai W, Anderson CS. Intracerebral haemorrhage: current approaches to acute management. Lancet. 2018 Oct 6;392(10154):1257-1268. doi: 10.1016/S0140-6736(18)31878-6. PMID 30319113
- [Result] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Result] Morgenstern LB, Hemphill JC 3rd, Anderson C, Becker K, Broderick JP, Connolly ES Jr, Greenberg SM, Huang JN, MacDonald RL, Messe SR, Mitchell PH, Selim M, Tamargo RJ; American Heart Association Stroke Council and Council on Cardiovascular Nursing. Guidelines for the management of spontaneous intracerebral hemorrhage: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2010 Sep;41(9):2108-29. doi: 10.1161/STR.0b013e3181ec611b. Epub 2010 Jul 22. PMID 20651276
- [Result] Mendelow AD, Gregson BA, Rowan EN, Murray GD, Gholkar A, Mitchell PM; STICH II Investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial lobar intracerebral haematomas (STICH II): a randomised trial. Lancet. 2013 Aug 3;382(9890):397-408. doi: 10.1016/S0140-6736(13)60986-1. Epub 2013 May 29. PMID 23726393
- [Result] Goyal N, Tsivgoulis G, Malhotra K, Katsanos AH, Pandhi A, Alsherbini KA, Chang JJ, Hoit D, Alexandrov AV, Elijovich L, Fiorella D, Nickele C, Arthur AS. Minimally invasive endoscopic hematoma evacuation vs best medical management for spontaneous basal-ganglia intracerebral hemorrhage. J Neurointerv Surg. 2019 Jun;11(6):579-583. doi: 10.1136/neurintsurg-2018-014447. Epub 2019 Jan 7. PMID 30617144
- [Result] Wang WZ, Jiang B, Liu HM, Li D, Lu CZ, Zhao YD, Sander JW. Minimally invasive craniopuncture therapy vs. conservative treatment for spontaneous intracerebral hemorrhage: results from a randomized clinical trial in China. Int J Stroke. 2009 Feb;4(1):11-6. doi: 10.1111/j.1747-4949.2009.00239.x. PMID 19236490
- [Result] Xia Z, Wu X, Li J, Liu Z, Chen F, Zhang L, Zhang H, Wan X, Cheng Q. Minimally Invasive Surgery is Superior to Conventional Craniotomy in Patients with Spontaneous Supratentorial Intracerebral Hemorrhage: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Jul;115:266-273. doi: 10.1016/j.wneu.2018.04.181. Epub 2018 May 3. PMID 29730105
- [Result] Lovelock CE, Molyneux AJ, Rothwell PM; Oxford Vascular Study. Change in incidence and aetiology of intracerebral haemorrhage in Oxfordshire, UK, between 1981 and 2006: a population-based study. Lancet Neurol. 2007 Jun;6(6):487-93. doi: 10.1016/S1474-4422(07)70107-2. PMID 17509483
- [Result] Baron TH, Kamath PS, McBane RD. Management of antithrombotic therapy in patients undergoing invasive procedures. N Engl J Med. 2013 May 30;368(22):2113-24. doi: 10.1056/NEJMra1206531. No abstract available. PMID 23718166
- [Result] Krittalak K, Sawanyawisuth K, Tiamkao S. Safety of withholding anticoagulation in patients with mechanical prosthetic valves and intracranial haemorrhage. Intern Med J. 2011 Oct;41(10):750-4. doi: 10.1111/j.1445-5994.2011.02579.x. PMID 22435901
- [Result] Cahill RA, McGreal GT, Crowe BH, Ryan DA, Manning BJ, Cahill MR, Redmond HP. Duration of increased bleeding tendency after cessation of aspirin therapy. J Am Coll Surg. 2005 Apr;200(4):564-73; quiz A59-61. doi: 10.1016/j.jamcollsurg.2004.11.002. PMID 15804471
- [Result] Korinth MC. Low-dose aspirin before intracranial surgery--results of a survey among neurosurgeons in Germany. Acta Neurochir (Wien). 2006 Nov;148(11):1189-96; discussion 1196. doi: 10.1007/s00701-006-0868-4. Epub 2006 Sep 21. PMID 16969624
- [Result] de Miguel-Diez J, Gomez Martinez A, Montero Martinez C. Perioperative and Periprocedural Management of Antithrombotic Therapy. Arch Bronconeumol (Engl Ed). 2019 May;55(5):229-230. doi: 10.1016/j.arbres.2018.07.019. Epub 2018 Sep 5. No abstract available. English, Spanish. PMID 30193947
- [Result] Douketis JD, Berger PB, Dunn AS, Jaffer AK, Spyropoulos AC, Becker RC, Ansell J. The perioperative management of antithrombotic therapy: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):299S-339S. doi: 10.1378/chest.08-0675. PMID 18574269
- [Result] Douketis JD, Bakhsh E. Perioperative management of antithrombotic therapy. Pol Arch Med Wewn. 2008 Apr;118(4):201-8. PMID 18575419
- [Result] Wijdicks EF, Schievink WI, Brown RD, Mullany CJ. The dilemma of discontinuation of anticoagulation therapy for patients with intracranial hemorrhage and mechanical heart valves. Neurosurgery. 1998 Apr;42(4):769-73. doi: 10.1097/00006123-199804000-00053. PMID 9574641
- [Result] Luddington RJ. Thrombelastography/thromboelastometry. Clin Lab Haematol. 2005 Apr;27(2):81-90. doi: 10.1111/j.1365-2257.2005.00681.x. PMID 15784122
- [Result] Kashuk JL, Moore EE, Sabel A, Barnett C, Haenel J, Le T, Pezold M, Lawrence J, Biffl WL, Cothren CC, Johnson JL. Rapid thrombelastography (r-TEG) identifies hypercoagulability and predicts thromboembolic events in surgical patients. Surgery. 2009 Oct;146(4):764-72; discussion 772-4. doi: 10.1016/j.surg.2009.06.054. PMID 19789037
- [Result] Naidech AM, Jovanovic B, Liebling S, Garg RK, Bassin SL, Bendok BR, Bernstein RA, Alberts MJ, Batjer HH. Reduced platelet activity is associated with early clot growth and worse 3-month outcome after intracerebral hemorrhage. Stroke. 2009 Jul;40(7):2398-401. doi: 10.1161/STROKEAHA.109.550939. Epub 2009 May 14. PMID 19443791
- [Result] Prasad K, Mendelow AD, Gregson B. Surgery for primary supratentorial intracerebral haemorrhage. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD000200. doi: 10.1002/14651858.CD000200.pub2. PMID 18843607
- [Result] Li Y, Yang R, Li Z, Yang Y, Tian B, Zhang X, Wang B, Lu D, Guo S, Man M, Yang Y, Luo T, Gao G, Li L. Surgical Evacuation of Spontaneous Supratentorial Lobar Intracerebral Hemorrhage: Comparison of Safety and Efficacy of Stereotactic Aspiration, Endoscopic Surgery, and Craniotomy. World Neurosurg. 2017 Sep;105:332-340. doi: 10.1016/j.wneu.2017.05.134. Epub 2017 May 31. PMID 28578111
- [Result] Yao Z, Ma L, You C, He M. Decompressive Craniectomy for Spontaneous Intracerebral Hemorrhage: A Systematic Review and Meta-analysis. World Neurosurg. 2018 Feb;110:121-128. doi: 10.1016/j.wneu.2017.10.167. Epub 2017 Nov 10. PMID 29129764
- [Result] Zheng J, Li H, Zhao HX, Guo R, Lin S, Dong W, Ma L, Fang Y, Tian M, Liu M, You C. Surgery for Patients With Spontaneous Deep Supratentorial Intracerebral Hemorrhage: A Retrospective Case-Control Study Using Propensity Score Matching. Medicine (Baltimore). 2016 Mar;95(11):e3024. doi: 10.1097/MD.0000000000003024. PMID 26986116
- [Result] Stein M, Misselwitz B, Hamann GF, Kolodziej M, Reinges MH, Uhl E. In-hospital mortality after pre-treatment with antiplatelet agents or oral anticoagulants and hematoma evacuation of intracerebral hematomas. J Clin Neurosci. 2016 Apr;26:42-5. doi: 10.1016/j.jocn.2015.05.069. Epub 2015 Dec 11. PMID 26690758
- [Result] Khoo KF, Lepas B. Summary of evidence-based guideline: Periprocedural management of antithrombotic medications in patients with ischemic cerebrovascular disease: report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2014 Jan 7;82(1):95. doi: 10.1212/01.NEUROLOGY.0000437348.92583.18. No abstract available. PMID 24379098
- [Result] Holzmacher JL, Reynolds C, Patel M, Maluso P, Holland S, Gamsky N, Moore H, Acquista E, Carrick M, Amdur R, Hancock H, Metzler M, Dunn J, Sarani B. Platelet transfusion does not improve outcomes in patients with brain injury on antiplatelet therapy. Brain Inj. 2018;32(3):325-330. doi: 10.1080/02699052.2018.1425804. Epub 2018 Jan 17. PMID 29341793
- [Result] Katz J, Feldman MA, Bass EB, Lubomski LH, Tielsch JM, Petty BG, Fleisher LA, Schein OD; Study of Medical Testing for Cataract Surgery Team. Risks and benefits of anticoagulant and antiplatelet medication use before cataract surgery. Ophthalmology. 2003 Sep;110(9):1784-8. doi: 10.1016/S0161-6420(03)00785-1. PMID 13129878